CLINICAL TRIAL: NCT06665022
Title: Neuromodulation Effects in Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been absorbed into a pre-existing, IRB-approved (IRB202202370) study with an active Clinical Trials page (NCT05998031). This IRB (IRB202401208) has been withdrawn.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB202401208
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Impairment; Cognitive Decline
Keywords: Cognitive Aging; Brain Stimulation; functional MRI; Computational Modeling; Finite Element Method (FEM)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will enroll in a randomized double-blinded crossover within subject study. Each participant will undergo two MRI sessions. Each MRI session will include either one active tDCS or one sham tDCS. The order of delivering active or sham tDCS first will be randomized. A washout period between active and sham tDCS will be set for at least two-weeks to ensure no after-effect from the first stimulation session will be carried over to the second session.
Who Masked: Participant, Outcomes Assessor
Masking Description: A blinding code will be entered into the stimulation device to initiate the randomized stimulation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): A neuroConn MR-safe 1x1 tDCS stimulator will be used to apply 12 minutes of 2.0 mA electrical current, with 30 seconds ramps up and 30 seconds ramps down. The electrical current will be applied by using two carbon rubber electrodes (one anode, one cathode) with added ten20 conductive paste. The electrode+paste will be affixed on the participant's scalp over the frontal cortices at F3 and F4 location (EEG 10-20 system). Inflow of current (anode) will occur at F4 location, and outflow of current will occur at F3 (cathode). For each stimulation condition (active, sham), each participant will perform two runs of N-back working memory task (baseline/pre-stimulation and during stimulation). Sham efficacy will be evaluated as a direct comparison in N-back performance and connectivity results in active group versus sham group.
  Interventions: Device: Active tDCS
- Sham tDCS (Placebo Comparator): Sham stimulation will be performed with the same 1x1 device. Participants will receive 2 mA of direct current stimulation for 30 seconds with 30 seconds ramps up and down. This provides the tingling and prickling sensation on the scalp associated with tDCS while prevent delivering sufficient current (12 minutes) to penetrate the skull and stimulate the brain. Prep in sham conditions will be identical to active stimulation conditions. For each stimulation condition (active, sham), each participant will perform two runs of N-back working memory task (baseline/pre-stimulation and during stimulation). Sham efficacy will be evaluated as a direct comparison in N-back performance and connectivity results in active group versus sham group.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — A neuroConn MR-safe 1x1 tDCS stimulator will be used to apply 12 minutes of 2.0 mA electrical current, with 30 seconds ramps up and 30 seconds ramps down. The electrical current will be applied by using two carbon rubber electrodes (one anode, one cathode) with added ten20 conductive paste. The electrode+paste will be affixed on the participant's scalp over the frontal cortices at F3 and F4 location (EEG 10-20 system). Inflow of current (anode) will occur at F4 location, and outflow of current will occur at F3 (cathode). For each stimulation condition (active, sham), each participant will perform two runs of N-back working memory task (baseline/pre-stimulation and during stimulation). Sham efficacy will be evaluated as a direct comparison in N-back performance and connectivity results in active group versus sham group.
  Arms: Active tDCS
Device: Sham tDCS — Sham stimulation will be performed with the same 1x1 device. Participants will receive 2 mA of direct current stimulation for 30 seconds with 30 seconds ramps up and down. This provides the tingling and prickling sensation on the scalp associated with tDCS while prevent delivering sufficient current (12 minutes) to penetrate the skull and stimulate the brain. Prep in sham conditions will be identical to active stimulation conditions. For each stimulation condition (active, sham), each participant will perform two runs of N-back working memory task (baseline/pre-stimulation and during stimulation). Sham efficacy will be evaluated as a direct comparison in N-back performance and connectivity results in active group versus sham group.
  Arms: Sham tDCS

SUMMARY:
The current study is a mechanistic study to evaluate working memory gains from application of transcranial direct current stimulation (tDCS) in older adults with mild cognitive impairments (MCI) compared to cognitively healthy control

DETAILED DESCRIPTION:
The current study is a mechanistic study to evaluate working memory gains with transcranial direct current stimulation (tDCS) in older adults with mild cognitive impairments (MCI) compared to cognitively healthy control. The proposed study investigates the effects of acute (one-time) tDCS application on working memory gains (i.e., behavior and functional) by evaluating brain structure and cognitive function relationships. tDCS is a method of non-invasive brain stimulation that directly stimulates brain regions involved in active cognitive function and enhances neural plasticity when paired with a training task. A mechanistic, in-scanner, crossover design tDCS study (active and sham stimulation) with 2milliamps (mA) fixed dosing application will enroll 110 participants comprising 55 cognitively normal/healthy older adults and 55 older adults with MCI. The study will employ multi-modal neuroimaging (structural and functional data), person-specific computational models, and machine learning to elucidate acute tDCS effects on working memory. Change in cognitive function (i.e., working memory performance) will be quantified using working memory tasks and magnetic resonance imaging (MRI). The investigators will compare changes in working memory performance resulting from active tDCS versus sham tDCS during 2-back task compared to 0-back task.

The investigators will test the following hypotheses:

1. Acute tDCS will increase working memory performance during active tDCS and larger degree of brain atrophy seen in MCI patients will significantly decrease current intensity in stimulated brain regions.
2. Acute tDCS will significantly increase functional connectivity within the working memory network during active tDCS but not sham.

The present study will provide insight into mechanisms underlying tDCS application in MCI population for combating cognitive decline in a rapidly aging population in the United States. Information gathered from this study may guide future intervention strategies to combat cognitive decline and improve the quality of life of aging population.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-95 years
* Montreal Cognitive Assessment (MoCA) score 18 and above (scores will be adjusted for education)
* Able to receive electrical stimulation
* Adequate motor capacity to participate in intervention and training sessions

Exclusion Criteria:

* Contraindications to MRI recording
* Left-handed
* Inability to communicate in English
* History of neurological/psychiatric disorders and traumatic brain injury
* Incidence of stroke
* Severe visual and hearing impairment precluding completion of study assessments

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
2-back Working Memory Accuracy | 12 minutes versus 24 minutes in each session. Then comparing active versus sham stimulation sessions, separated by at least two weeks.
  The descriptive name of the scale is 2-back Working Memory Accuracy. Participants will perform in-scanner 0 and 2-back (i.e., N-back) working memory task that asks them to acknowledge whether a letter was the same as the letter 2 or N times before. Participant will view one letter at a time, with a crosshair appear briefly as an inter-stimulus interval. The task paradigm for each run consists of four blocks of 2-back and four blocks of 0-back. Two runs (before and during stimulation) will be performed at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Aprinda I Queen, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States